CLINICAL TRIAL: NCT06835894
Title: Do End-Tidal Capnography Trends Reflect Changes in Arterial Carbon Dioxide Partial Pressure During One-Lung Ventilation for Thoracoscopic Surgery? A Prospective Observational Study
Brief Title: Trending Ability of End-Tidal Capnography to Reflect Arterial Carbon Dioxide Changes in One-Lung Ventilation
Status: Not yet recruiting | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Kamil Darcin, Associate Professor, Koç University
Other Study IDs: 2024.269.IRB1.033
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Video-Assisted Thoracoscopic Surgery; One-Lung Ventilation; Capnography; Blood Gas Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we want to find out if measuring carbon dioxide from a patient's breath (end-tidal CO₂ or ETCO₂) can reliably reflect changes in blood carbon dioxide levels (arterial CO₂ or PaCO₂) during lung surgery. Instead of just looking at individual values, we are specifically investigating whether ETCO₂ and PaCO₂ rise and fall in the same direction over time.

During lung surgery, patients often need "one-lung ventilation," where only one lung is used for breathing while the other is deflated to help the surgeon. This can cause carbon dioxide levels in the blood to change, which are typically monitored by taking blood samples. If ETCO₂ trends closely follow PaCO₂ trends, doctors may not need to take as many blood samples.

Patients in this study will already have a small tube in an artery for monitoring blood pressure. Whenever a blood test is taken, we will compare the blood CO₂ level with the ETCO₂ reading at that moment. We will also track heart rate, blood pressure, and body temperature.

By comparing these measurements, we hope to learn whether ETCO₂ reliably follows the same trends as PaCO₂, making it a useful tool for monitoring carbon dioxide levels in lung surgery with fewer blood tests.

DETAILED DESCRIPTION:
Thoracoscopic lung surgery often requires one-lung ventilation, a technique in which only one lung is ventilated while the other is deflated to provide better access for the surgeon. This can lead to changes in blood carbon dioxide (PaCO₂) levels, which must be monitored closely to ensure patient safety. Arterial blood gas sampling remains the gold standard for measuring PaCO₂, but it is invasive, costly, and provides only intermittent data. End-tidal carbon dioxide (ETCO₂) monitoring, available through standard anesthesia devices, offers continuous, noninvasive measurement of exhaled CO₂ and can serve as a surrogate for PaCO₂.

The primary purpose of this study is to evaluate the agreement and trend correlation between ETCO₂ and PaCO₂ in patients undergoing thoracoscopic procedures with one-lung ventilation. If ETCO₂ reliably tracks changes in PaCO₂, clinicians may reduce the number of arterial blood gas samples required during these operations.

Primary objective: To evaluate the trend correlation between ETCO₂ and PaCO₂ over time.

Secondary objective: To determine the degree of agreement between ETCO₂ and PaCO₂

Study Type: Prospective, observational study. Study Setting: Operating rooms where adult patients (≥18 years old) are scheduled for thoracoscopic procedures with one-lung ventilation and require invasive arterial pressure monitoring as part of their routine care.

Duration: Each patient's participation will be limited to the intraoperative period (i.e., from anesthesia induction to the end of surgery).

Intraoperative management will follow a standardized anesthetic protocol, and arterial blood gas samples will be drawn at the anesthesiologist's discretion whenever clinically indicated.

Each time an arterial blood gas sample is taken, the corresponding ETCO₂, PaCO₂, arterial blood pressure, heart rate, and temperature values will be recorded.

Any use of inotropic or antihypertensive infusions will be documented, as such medications can influence hemodynamic stability and possibly ventilatory parameters.

The patient's demographic details (age, sex, height, weight) and the type of surgical procedure will be recorded.

Four-quadrant plots will be generated to assess the concordance of changes in ETCO₂ with changes in PaCO₂ over time.

Bland-Altman plots will be constructed to calculate the mean difference (bias) and 95% limits of agreement for each paired measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracoscopic lung surgery with one-lung ventilation
* Patients requiring invasive arterial blood pressure monitoring

Exclusion Criteria:

* Chronic obstructive pulmonary disease (COPD)
* Pulmonary hypertension
* Systemic infection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be drawn from the adult patient population (≥18 years) scheduled for thoracoscopic lung surgery with one-lung ventilation at a tertiary care hospital. These individuals are already indicated to receive invasive arterial blood pressure monitoring as part of their routine clinical management. No special outreach or community recruitment methods will be employed; rather, eligible patients will be identified from the hospital's surgical wards and preoperative clinics.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Trend correlation between ETCO₂ and PaCO₂ measured by the concordance ratio in the four-quadrant plot | During the surgery of the patient, arterial blood gas samples will be drawn at the anesthesiologist's discretion whenever clinically indicated.
  A four-quadrant plot will be generated by comparing consecutive changes (deltas) in PaCO₂ and ETCO₂. For each patient, every pair of sequential measurements will be used to calculate ΔPaCO₂ (horizontal axis) and ΔETCO₂ (vertical axis). Points in the top-right (Quadrant I) and bottom-left (Quadrant III) indicate concordant changes (both variables increased or both decreased). A "central zone" will be defined to exclude clinically negligible fluctuations (±1mmHg). The percentage of points in Quadrant I and III, relative to those outside the central zone, will be reported as the overall concordance. A concordance ratio above 90% will be considered as good trending ability.
Trend correlation between ETCO₂ and PaCO₂ measured by the angular bias in the four-quadrant plot | During the surgery of the patient, arterial blood gas samples will be drawn at the anesthesiologist's discretion whenever clinically indicated.
  In the four-quadrant plot, the angle of each data point relative to the 45-degree line will be calculated. The average of this angles will be reported as angular bias. An angular bias between ±5 degrees will be considered as good trending ability.
Trend correlation between ETCO₂ and PaCO₂ measured by radial limits of aggreement in the four-quadrant plot | During the surgery of the patient, arterial blood gas samples will be drawn at the anesthesiologist's discretion whenever clinically indicated.
  In the four-quadrant plot, the angle of each data point relative to the 45-degree line will be calculated. The radial sector relative to the 45-degree line that contains 95% of the data points will be reported as radial limits of agreement. Radial limits of agreement between ±30 degrees will be considered as good trending ability.

SECONDARY OUTCOMES:
Aggreement between simultaneous ETCO₂ and PaCO₂ values measured by limits of aggreement in Bland-Altman plot | During the surgery of the patient, arterial blood gas samples will be drawn at the anesthesiologist's discretion whenever clinically indicated.
  A Bland-Altman plot will be used to assess agreement between ETCO₂ and PaCO₂. For each paired measurement, the difference between ETCO₂ and PaCO₂, and the average of ETCO₂ and PaCO₂ will be calculated. Each point will be plotted with the difference on the vertical axis against the average on the horizontal axis. The mean difference (bias) and 95% limits of agreement (mean difference ± 1.96 × Standard deviation of the difference) will then be calculated. Limits of aggreement between ±4 mmHg will be considered as good aggreement.